CLINICAL TRIAL: NCT03437356
Title: Pulmonary Vein Isolation With Versus Without Continued Antiarrhythmic Drug Treatment in Subjects With Persistent Atrial Fibrillation: a Prospective Multi-centre Randomized Controlled Clinical Study
Brief Title: Pulmonary Vein Isolation With Versus Without Continued Antiarrhythmic Drugs in Persistent Atrial Fibrillation
Acronym: POWDER-AF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Mattias Duytschaever, Prof. Dr., AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8049201834825
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: persistent atrial fibrillation; pulmonary vein isolation; antiarrhythmic drug therapy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT ON Group (Active Comparator): 'CLOSE'-guided PVI with continuation of antiarrhythmic drug therapy (ADT) at the end of the 3-months blanking period after ablation.
  Interventions: Other: Pulmonary vein isolation using CLOSE protocol; Drug: Antiarrhythmic drug therapy (ADT)
- ADT OFF Group (Active Comparator): 'CLOSE' guided PVI with discontinuation of antiarrhythmic drug therapy (ADT) at the end of the 3-months blanking period after ablation
  Interventions: Other: Pulmonary vein isolation using CLOSE protocol

INTERVENTIONS:
Other: Pulmonary vein isolation using CLOSE protocol — 'CLOSE' protocol: Ablation index > 400 at the posterior wall (reduce to 300 if esophagus temperature rise), ablation index > 550 at the anterior wall, and inter-lesion distance < 6.0mm
Drug: Antiarrhythmic drug therapy (ADT) — During the first 3 months after PVI, patients continue oral anticoagulants and antiarrhythmic drug therapy (ADT). ADT is a continuation (or restart) of previously ineffective Class IC and III ADT. At the time of discharge, dosage is optimized according to the 2016 ESC guidelines on AF management.
  Preferred dosages:
  Flecainide: Tambocor or Flecainide EG 100mg b.i.d., Apocard R 100 to 200mg overdose (OD) Propafenone: Rytmonorm or Propafenone EG 300 mg b.i.d., except 225 mg b.i.d. if ≥70 years or <70 kg Sotalol: Sotalex or Sotalol EG 80mg b.i.d., Except 80mg t.i.d. if men < 70 years, Cr <1.5mg/dl, >70kg, except 80 mg OD if female >70 years or Cr >1.2mg/dl
  In case of amiodarone intake before PVI, amiodarone is switched to sotalol or class IC ADT.
  Arms: ADT ON Group

SUMMARY:
In the POWDER 1 study, paroxysmal atrial fibrillation (AF) patients undergoing conventional contact force (CF)-guided PVI were investigated. Patients were randomized between continuing previously ineffective antiarrhythmic drug therapy (ADT) or stopping ADT at the end of the blanking period. This trial, showed an added value of ADT after ablation (in support of 'hybrid rhythm control' as an alternative treatment strategy for AF in some patients).

In the POWDER 2 trial, an analogue study in persistent AF patients will be performed. All patients will undergo ablation index (AI)- and IL distance (ILD)-guided PVI (just like in VISTAX trial) and continue previously ineffective ADT during the blanking period. 'PVI only' was chosen as the ablation strategy according to the STAR AF trial findings.

DETAILED DESCRIPTION:
Background: In real-life, ADT is often continued after catheter ablation for persistent AF. No study investigated whether ADT continued beyond the blanking period reduces recurrence after a first ablation for persistent AF.

Purpose: The aim of this trial is to investigate whether continued ADT (ADT ON) reduces recurrence of atrial tachyarrhythmia (ATA) in the first year after contact-force guided PVI for persistent AF.

Hypothesis: Continued use of ADT beyond the blanking period reduces recurrence of ATA in the first year after PVI .

Eligibility: Subjects that are planned for catheter ablation for persistent AF.

Inclusion: Symptomatic persistent AF resistant to ongoing or prior ADT (failed ADT). Persistent AF is defined as the presence of any prior AF episode ≥7 days.

Exclusion: Any prior AF episode ≥12 months, any recurrence of AF <3 days after cardioversion.

Echo criteria: advanced valvular heart disease, left atrium (LA) volume >37ml/m2, left ventricle (LV) ejection fraction <35% (except if suspected tachycardiomyopathy), septal diameter >15mm, Life expectancy <1 year, BMI >35.

Trial design: This is a prospective, multi-center, randomized (1:1), open label, blinded endpoint study (PROBE). Eligible subjects who sign the study informed consent form at the time of procedural planning will be randomized into one of two study arms: In the ADT off arm (ADT OFF), ADT will be stopped at 3 months after the first procedure. In the ADT ON arm, ADT will be continued at 3 months until 1 year follow up (FU).

First ablation and blanking: In both arms, catheter ablation will consist of 'CLOSE'-guided PVI only (abl index and interlesion distance). High-density voltage mapping will be performed during sinus rhythm. After ablation, ADT is continued/restarted during the 3-month blanking period (except for amiodarone). During the blanking period cardioversions are allowed. At the 3-month visit, all patients will be cardioverted if ATA is present.

Repeat ablation strategy: In case of recurrence of ATA's after 3 months, a repeat ablation is recommended. Depending on the reconnection status of the pulmonary veins (PV), repeat ablation will consist of either PVI only or a patient-tailored ablation approach (antral isolation, superior vena cava (SVC) isolation, isolation of low voltage, linear lesions). Patients stay on the ADT ON or ADT OFF arm.

Primary Endpoint: Any documented ATA (atrial fibrillation, AF, atrial tachycardia, AT, atrial flutter, AFL) lasting >30s from 3 months through 12 month follow-up after the first procedure.

Secondary Endpoints:

ATA recurrence in patients with early peristent AF (defined as AF ≤3 months) Incidence of repeat ablation Unscheduled visits and hospitalisation ADT or ablation related adverse events QOL and symptoms Outcome after repeat ablation

Sample size: In the ADT OFF group ATA recurrence after a first PVI is expected to be 50%. ADT are expected to reduce ATA recurrence to 30%. Given power of 80% and α of 0.05 up to 200 subjects need be enrolled in this study (20 per center)

ELIGIBILITY:
Inclusion Criteria:

1. Patient with symptomatic persistent AF, resistant to ongoing or prior ADT (failed ADT) Patients is considered to have persistent AF if the patient has suffered any prior AF episode ≥7 days (ESC 2016 guidelines).
2. Before PVI, there was at least one episode of persistent AF in the last year.
3. Signed Patient Informed Consent Form.
4. Age 18 years or older.
5. Able and willing to comply with all follow-up testing and requirements.

Exclusion Criteria:

1. Patients not willing or not suited to take any class IC or III ADT.
2. Any prior AF episode ≥12 months, or any recurrence of AF <3 days after cardioversion.
3. Presence of structural heart disease on echo criteria:

   severe valvular heart disease; LA diameter >50mm; LV ejection fraction <35% (except if suspected tachycardiomyopathy); septal diameter >15mm
4. BMI >35
5. Recent (<3 months) coronary artery bypass grafting (CABG), myocardial infarction, cerebral vascular accident (CVA), uncontrolled heart failure or angina
6. Active illness or systemic infection or sepsis
7. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
8. Awaiting cardiac transplantation or other cardiac surgery
9. Documented left atrial thrombus or atrial myxoma on imaging
10. History of blood clotting or bleeding abnormalities
11. Enrollment in any other study evaluating another device or drug
12. Women with childbearing potential
13. Life expectancy less than 12 months
14. Contraindication for catheter ablation (intramural thrombus, tumor or other abnormality that precludes catheter introduction, contraindication to anticoagulation therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Any documented AF/atrial tachycardia (AT)/atrial flutter (AFL) recurrence | From 3 to 12 months after PVI
  Recurrence will be considered as AF/AT/AF lasting >30 seconds, as measured by 1-day Holter monitoring at 6 month after PVI, 7-day Holter (screening for AF between 48 hours and 7 days) at 12 months after PVI, and by any standard of care or unscheduled arrhythmia monitoring documentation throughout the follow-up (ie. from 3 to 12 months after PVI).

SECONDARY OUTCOMES:
AF/atrial tachycardia (AT)/atrial flutter (AFL) recurrence in early persistent AF | From 3 to 12 months after PVI
  Incidence of recurrence of early persistent AF
Repeat ablation | From 3 to 12 months after PVI
  Incidence of repeat ablation
Unscheduled health care visits and hospitalizations | From 3 to 12 months after PVI
  Incidence of unscheduled health care visits and/or hospitalizations
ADT-related adverse events | From 3 to 12 months after PVI
  Adverse events related to continuation of ADT in the ON group
Ablation-related adverse events | From 0 to 12 months after ablation
  Adverse events related to ablation in both groups
Quality of life assessment (SF-36) | At Enrollment, and at 3 months, 6 months, and 12 months after ablation
  At each scheduled visit, the patients will fill the SF-36 questionnaire for the assessment of Quality of life before and after ablation in both groups. SF-36 individual scores (0-100) will be converted into z-scores as standardized combined scores (mean 50, standard deviation 10) for US population (Ware et al.)
AF symptom scores | At Enrollment, and at 3 months, 6 months, and 12 months after ablation
  At each scheduled visit, the patients will fill AF checklist: 16 questions of AF severity (score = minimum 16, maximum 48) and 16 questions of AF frequency (score = minimum 16, maximum 64) for qualitative assessment of AF symptoms before and after ablation in both groups.
Predictors of recurrence | At baseline
  Any conventional clinical characteristics acquired at baseline that could predict recurrence of AF
Outcome after repeat ablation | From 3 to 12 months after first PVI
  Incidence of AF recurrence after multiple ablation procedures (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Duytschaever, MD, PhD, Principal Investigator — A Sint -Jan Bruges
Locations (9):
- Medical University of Graz, Graz, Austria
- Belgium (5):
  - Onze-Lieve-Vrouwziekenhuis Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan Hospital, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis Hasselt, Hasselt
- Gentofte Hospital, Gentofte Municipality, Denmark
- Hospital Universitari Germans Trias, Barcelona, Spain
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demolder A, O'Neill L, El Haddad M, Scherr D, Vijgen J, Wolf M, Berte B, Bisbal F, Johannessen A, Rivero-Ayerza M, De Potter T, De Becker B, Polain de Waroux JL, Knecht S, Tavernier R, Duytschaever M. No Effect of Continued Antiarrhythmic Drug Treatment on Top of Optimized Pulmonary Vein Isolation in Patients With Persistent Atrial Fibrillation: Results From the POWDER-AF2 Trial. Circ Arrhythm Electrophysiol. 2023 Nov;16(11):e012043. doi: 10.1161/CIRCEP.123.012043. Epub 2023 Nov 3. PMID 37921006